CLINICAL TRIAL: NCT07185529
Title: Predictors of Mortality in Multiple Trauma Patients With Intensive Care Unit: A Retrospective Cohort Study
Brief Title: Predictors of Mortality in Multiple Trauma Patients
Status: Completed | Type: Observational
Sponsor: Melike Cengiz (Other)
Responsible Party: Sponsor-Investigator, Melike Cengiz, professor doctor, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: Akdeniz.
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Multiple Trauma/Injuries
Keywords: Intensive Care Unit; Mortality; Multiple trauma patient
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- survival: consists of surviving patients
  Interventions: Other: Data of the patients were obtained from patient observation files and hospital information system database.
- mortality: consists of deceased patients
  Interventions: Other: Data of the patients were obtained from patient observation files and hospital information system database.

INTERVENTIONS:
Other: Data of the patients were obtained from patient observation files and hospital information system database. — Data of the patients were obtained from patient observation files and hospital information system database.

SUMMARY:
Trauma is a public health concern that causes serious financial and medical burdens worldwide. According to the World Health Organization, 4.4 million people die from traumatic injuries each year which account for about 8% of global deaths. Traumatic injuries are among the most common causes of mortality particularly in young individuals. It also has a negative economic impact due to the loss of labor. Determining the factors associated with mortality in the ICU follow-up and treatment of these patients is very important for clarifying these uncertainties and improving ICU outcomes. The main objective of the study was to ascertain the ICU processes of multipletrauma patients and the factors that may have an effect on mortality.

DETAILED DESCRIPTION:
All patients with traumatic injuries severe enough to warrant ICU admission formed the subjects of the study. The study included patients aged 18 years and over who were diagnosed with multiple trauma injuries and admitted to the ICU.The analysis included patients with a final outcome (survival or death) at our centre. Only patients who were admitted to the ICU for the first time were included. The following systems were used to assess the clinical and multiple trauma injury severity at the time of admission to the ICU: the Acute Physiology and Chronic Health Assessment II (APACHE II) score, the Simplified Acute Physiology Score II (SAPS II), the Sequential Organ Failure Assessment (SOFA) score, the Glasgow Coma Scale (GCS), the Injury Severity Score (ISS), the Revised Trauma Score (RTS) and the Trauma and Injury Severity Score (TRISS). All injury severity scores were calculated using clinical findings, imaging results and surgical findings. A comprehensive data set was collated at the time of admission to the intensive care unit, encompassing patient age, gender, comorbidities, and the Charlson Comorbidity Index (CCI). The injury mechanism, blood sugar, haemoglobin and lactate levels, Horowitz index, hypotension and hypothermia were also recorded.The patients were categorised into two groups: survival and mortality

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with patients with multiple trauma injuries
* Patients with a final outcome (survival or mortality) in our centre

Exclusion Criteria:

* Patients with trauma to a single region (head, thorax, abdomen or extremities)
* Patients who were pregnant
* Length of intensive care unit stay ≤24 hours

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The sample included patients with multiple trauma injuries who were admitted in the ICU between 01 January 2021 and 01 November 2023.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is mortality | 01 January 2021 and 01 November 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)